CLINICAL TRIAL: NCT05943249
Title: Development of Novel MR Techniques Using Volunteer Participants
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 3T000175
Record Dates: First submitted 2023-06-26; First posted 2023-07-13 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Healthy
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: magnetic resonance

SUMMARY:
Using magnetic resonance (MR) imaging or spectroscopy as part of clinical research typically involves developing new MR protocols. Although some of this work is done by scanning artificial 'phantoms', volunteer studies are normally needed to configure and validate new protocols appropriately.

Developing new MR protocols and techniques is also useful in its own right. The volunteer scanning described in this application will provide data to support this type of methodological research into new scanning and image processing techniques: improving the speed, quality, and range of measurements possible with the scanner.

With proper safety and screening procedures, MR has no known side-effects, and has been performed on millions of human subjects worldwide without ill effect. There are well-established contraindications for MRI, and screening procedures are already in place in the MR unit at UCLH to exclude such subjects and ensure the safety of subjects. With these, and the MR scanner's built in safety mechanisms, residual risk is low. Many other trusts with active MR research have previously made similar applications to this related to volunteer MR scanning for pilot work and methodological research

Although scans may obtained as part of several research projects, in each case it is only the scanning technique (the programmed sequence of data acquisition and processing steps) which will vary, along with the body region to be imaged. The volunteer experience will be very similar, and all ethical issues, including the information sheet and consent form, will be identical. These scans are for methodological research on the MR techniques themselves, and will be never form part of the volunteer's own healthcare. Separate ethical permission is sought for any study which does not match the above criteria.

DETAILED DESCRIPTION:
We are applying for general permission to acquire magnetic resonance (MR) data from normal volunteers. Data will be used to develop and test MR protocols for subsequent clinical research, and to support methodological research into MR techniques: improving the speed, quality, and range of measurements possible with the scanner. This application is restricted to the non-invasive imaging of healthy adults. It excludes interventional MR procedures, injections of MR contrast agents, and all other invasive techniques. MR imaging has been performed on millions of subjects worldwide without ill effect: there are well-established contraindications for MR, particularly associated with metal in the body, and when these are followed residual risk is low. Scans will be performed on commercially available MR systems at UCLH, with their internal monitoring and safety devices always enabled. Scans will be connected with several research projects, but in each case it is the scanning technique (the programmed sequence of data acquisition and processing steps) which will vary. The volunteer experience will be similar, and all ethical and consent details will be identical. These scans are for methodological research on the MR techniques themselves, and will never form part of the volunteer's own healthcare. Volunteers will normally be recruited from within the medical physics department. Before scanning, the volunteer will undergo safety screening (a questionnaire, backed up by explanation from an MR radiographer or experienced MR physicist). If there are no contraindications to the scan, the volunteer will then be placed on a table inside the MR scanner. Ear protection will be provided. Occasionally, small temporary surface makers (usually ordinary cod liver oil capsules) may be placed on the volunteer's skin to allow positions to be identified between scans. Appropriate MR coils (receivers in plastic moldings, connected to the scanner by a cable) will usually be placed around the body part being imaged. Imaging will be carried out for a variable period of time not exceeding two hours. During the procedure, the volunteer may sometimes be asked to hold their breath or move in certain ways. Microphones, speakers, and an emergency buzzer allow the volunteer to remain in verbal contact with the person operating the scanner, and to request that the scan be terminated at any time for any reason. Normally, individual scans are independent. Occasionally a volunteer may be asked in advance to attend for more than one scan, to check that a newly designed measurement is reproducible across different visits. (It is anticipated, however, that some individuals will volunteer for several independent scans.)

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers will be recruited by email from within departments at UCL and UCLH
* male or female
* Aged 18 and above

Exclusion Criteria:

* volunteers with pacemakers or other implanted devices, or with other metallic foreign bodies, will be excluded.
* Women who may be pregnant
* any participants who cannot give informed consent (including anyone who may not adequately understand the verbal explanations or written information given in English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participant with the relevant condition Participant without condition Pre-condition Professionals Carers Relations Other Diagnostic, screening or prevention participants Genetically predisposed
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2007-06-04 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Development of novel MR techniques | 1 year
  New protocols will be developed and validated to be used in clinical research, and to provide volunteer data for ongoing research into magnetic resonance techniques: improving the speed, quality, and range of measurements possible with the scanner.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT05943249/Prot_000.pdf
  • Informed Consent Form (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT05943249/ICF_001.pdf